CLINICAL TRIAL: NCT04855214
Title: Patient-specific Requirements and Experiences of Upper Limb Prosthetic Technology
Brief Title: Evaluating the Experience of Upper Limb Prosthesis Use
Status: Recruiting | Type: Observational
Sponsor: Louis Stokes VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emily Graczyk, Career Scientist, Louis Stokes VA Medical Center
Other Study IDs: 20-02
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Prosthesis User; Amputation; Upper Limb Amputation at the Wrist; Upper Limb Amputation Above Elbow (Injury); Upper Limb Amputation Below Elbow (Injury)
Keywords: Upper Limb Prosthesis User; Survey; Interview; User Experience; Body-powered; Myoelectric; Multiple degree of freedom; Sensory Feedback; Prosthetic device features; Upper Limb Loss; Amputee; Outcome Acceptance; Qualitative Research
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Body-powered Prosthesis User: Individuals who use a prosthesis that relies on a system of cables or harnesses which are operated using other parts of the body like the shoulders, chest, or elbows.
  Interventions: Other: Qualitative Analysis
- Single degree-of-freedom (DOF) myoelectric prosthesis users: Individuals who use a myoelectric prosthesis that can perform only one movement.
  Interventions: Other: Qualitative Analysis
- Multi-DOF myoelectric prosthesis users: Individuals who use a myoelectric prosthesis that can perform more than one movement.
  Interventions: Other: Qualitative Analysis
- Sensory Augmentation: Individuals who experience augmented prosthesis sensory feedback through vibrating devices or pressure bladders, using electrical stimulation applied to the residual limb, or using neural implants.
  Interventions: Other: Qualitative Analysis

INTERVENTIONS:
Other: Qualitative Analysis — Mixed methods analysis of the user's experience with upper limb prosthetics.
  Other Names: Mixed Methods

SUMMARY:
The goal is to understand the critical factors associated with outcome acceptance following upper limb loss. The investigators aim to develop a unified theoretical model that describes the psychosocial experience of upper limb prosthesis use and predicts outcome acceptance following upper limb loss. The investigators will also examine experiences with prosthesis education, selection, and training as well as how psychological and social issues impact prosthesis use. In addition, the investigators will use the findings to develop a prototype decision tool to assist with matching persons to prostheses. Study findings will help providers, technology developers, and researchers better understand the complex experience of upper limb prosthesis use.

This conceptual framework will enable clinicians and researchers to evaluate and predict patient outcomes following limb loss, and to design interventions that improve outcomes. The proposed study is a mixed methods (qualitative and quantitative) study using an observational design. The qualitative component of the study will involve data collection through telephone interviews with 42 participants and analyses using a grounded theory approach with constant comparison methods. The quantitative component involves administration of standardized measures quantifying constructs of the theoretical model in 120 participants and analyses to produce a structural equation model of outcome acceptance. Participants will include persons with unilateral acquired upper limb loss at the trans radial or trans humeral level who use currently available prosthetic devices. Up to 16 individuals will participate in a series of focus groups that will be conducted to provide feedback on the model generated from previous data.

DETAILED DESCRIPTION:
Background Use of an upper limb prosthesis can improve function and quality of life, but these devices are frequently abandoned or used only intermittently. Two critical reasons for abandonment identified by prosthesis rejecters are insufficient prosthesis functionality and insufficient sensory feedback. Living with major limb loss is a complex experience involving multiple physical, psychological, and social factors. While many studies have investigated the needs and design priorities of prosthesis users, few have investigated how prosthesis features interact with other psychosocial aspects of the prosthesis use experience and overall attitude towards or acceptance of the device (outcome acceptance). To provide better prosthetic device options and improve rehabilitation outcomes, investigators must understand the relationships between prosthesis functional and sensory capabilities, the subjective experience of the prosthesis, and outcome acceptance following limb loss.

Objective The goal is to understand the critical factors associated with outcome acceptance following upper limb loss. The investigators aim to develop a unified theoretical model that describes the psychosocial experience of upper limb prosthesis use and predicts outcome acceptance following upper limb loss. This conceptual framework will enable clinicians and researchers to evaluate and predict patient outcomes following limb loss, and to design interventions that improve outcomes.

Specific Aims Aim 1: Assess the impact of the experience of prosthesis dexterity and control on outcome acceptance. Aim 2: Assess the impact of sensory feedback experience on outcome acceptance. Aim 3: Refine the theoretical model derived from qualitative analyses by exploring the quantitative relationships between aspects of the model of outcome acceptance. Aim 4: Examine how access to care and experiences with care shape acceptance of prosthetic devices Aim 5: Examine how perceived societal views affect prosthesis choice and acceptance Aim 6: Examine how patient-specific needs interact with expectations about device benefits and limitations to impact prosthesis acceptance Aim 7: Utilize clinician input and findings from qualitative analyses to design a prototype decision tool (TOP-MATCH) to facilitate matching patients with upper limb prostheses

Hypotheses For aims 1-3: Qualitative analyses will yield a theoretical model of outcome acceptance that includes psychosocial factors and prosthetic device factors related to dexterity, control, and sensory feedback. We hypothesize that experiences of prosthesis dexterity, control, and sensory feedback will both directly influence and modulate psychosocial factors of prosthesis use and user attitudes. We hypothesize that quantitative data collected through survey research will triangulate findings from the qualitative analyses, confirm the directionality of the conceptual relationships, and predict the relative weightings of relationships.

For aims 4-7: The long-term goal of this line of research is to improve satisfaction with and adoption of upper limb prostheses. The overarching objectives of this proposal are to 1) produce a grounded theory explaining how patient-specific needs, expectations, psychosocial factors, and care experiences interact with prosthetic device features to drive prosthesis acceptance and 2) use this framework to develop a prototype decision tool to assist with matching persons to prostheses. The theoretical model will help providers, technology developers, and researchers better understand the complex experience of upper limb prosthesis use. The clinical decision tool will incorporate the theoretical model to help clinicians and researchers navigate patient-specific needs and preferences to better optimize patient-specific technology prescription and identify best approaches to mitigate device abandonment. The research findings will be useful for increasing prosthesis satisfaction and decreasing rejection rates, ultimately helping providers and health systems make decisions to utilize resources judiciously.

Study Design The proposed study is a mixed methods (qualitative and quantitative) study using an observational design. The qualitative component of the study will involve data collection through telephone interviews with 42 participants and analyses using a grounded theory approach with constant comparison methods. The quantitative component involves administration and analyses of standardized measures quantifying constructs of the theoretical model in 120 participants and use of these measures in a structural equation model of outcome acceptance. Participants will include persons with unilateral acquired upper limb loss at the trans radial or trans humeral level who use currently available prosthetic devices. Using the above information, 16 individuals will participate in a series of focus groups that will be conducted to provide feedback on the model created.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Ability to give verbal informed consent
* Ability to speak and understand English
* Unilateral acquired trans-radial or trans-humeral amputee
* At least six months from time of limb loss
* Current user of an upper limb prosthesis
* Use of the device they will be describing for at least six months (with the exception of sensory augmentation)

Exclusion Criteria:

* Significant hearing impairment which would prevent telephone communication.
* Unwillingness or inability to discuss experiences with prostheses
* Emotional disturbance related to discussion the prosthesis or limb loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The proposed study will recruit a total of 138 persons with unilateral upper limb loss at the trans radial or trans humeral level. Participants may be users of any currently available prosthetic device brand, model, or terminal device, as long as their prosthesis can be classified into one of the four groups : 1) body-powered prosthesis users, 2) single degree-of-freedom (DOF) myoelectric prosthesis users, 3) multi-DOF myoelectric prosthesis users, and 4) user's who experience augmented sensory feedback in their prosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Estimated)
Dates: Start 2020-12-16 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient Experience Measure (PEM) | Two years
  Measures the participant's perception of various psychosocial outcomes including self-efficacy, embodiment, body image, prosthesis efficiency, and social touch. It is rated 0-4, where a higher score in each sub-scale indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Emily L Graczyk, PhD, Principal Investigator — Louis Stokes VA Medical Center; Dustin J Tyler, PhD, Principal Investigator — Louis Stokes VA Medical Center
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data will be made available upon request.